CLINICAL TRIAL: NCT00249197
Title: A Multicenter, Randomized, Open-Label Study to Compare the Safety and Efficacy of i.v. And/Or Oral Levofloxacin With That of Ticarcillin/Clavulanate Alone or Followed by Amoxicillin/Clavulanate in the Treatment of Complicated Bacterial Skin and Skin Structure Infections
Brief Title: A Study of the Safety and Effectiveness of Levofloxacin Compared to Ticarcillin/Clavulanate Alone or Followed by Amoxicillin/Clavulanate in the Treatment of Complicated Skin Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005473
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-01

CONDITIONS: Skin Diseases, Bacterial
Keywords: skin infection; bacterial infection; levofloxacin; quinolones; skin; infection
MeSH Terms: conditions — Skin Diseases, Bacterial; Cellulitis; Bacterial Infections; Infections | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of levofloxacin (an antibiotic) with ticarcillin/clavulanate alone or followed by amoxicillin/clavulanate in the treatment of complicated skin infections.

DETAILED DESCRIPTION:
Levofloxacin is an antibiotic that has been evaluated in clinical trials for use in the treatment of many types of infections including respiratory tract, urinary tract, and uncomplicated skin infections. Levofloxacin may be taken by mouth or administered slowly through a vein and has been shown to be safe and effective when administered once daily. This multicenter, open-label study will evaluate the safety and effectiveness of a single daily oral or intravenous dose of levofloxacin compared to multiple daily intravenous doses with another antibiotic, ticarcillin/clavulanate given alone or followed by oral amoxicillin/clavulanate, in the treatment of bacterial skin infections. Patients will receive 750 mg of levofloxacin by mouth or intravenously for 7 - 14 days, or 3.1 grams of ticarcillin/clavulanate intravenously for 7 - 14 days. Patients receiving levofloxacin intravenously may be switched to receive levofloxacin by mouth; patients receiving ticarcillin/clavulanate intravenously may be switched to 875 mg of amoxicillin/clavulanate given by mouth, twice daily, if significant improvement is noted. Patients are assessed after 3 - 4 days of treatment; treatment is discontinued if no significant improvement is noted. Patients showing signs of improvement continue in the study, with assessments 2 - 5 days (post-therapy visit) and 3 - 4 weeks (post-study visit) after completion of the study drug. The primary measure of effectiveness is the clinical response rate assessed 2 - 5 days after the last dose of antibiotic treatment, categorizing the response as cured, improved, or failed. Laboratory tests for the presence of bacteria are performed throughout the study. Safety evaluations (incidence of adverse events, physical examinations, laboratory tests) are performed throughout the study. The study hypothesis is that a single daily dose of levofloxacin is at least as effective as multiple daily doses of ticarcillin/clavulanate alone or followed by amoxicillin/clavulanate in the treatment of skin infections, and that it is well tolerated. Levofloxacin 750 mg intravenously or by mouth, once daily for 7 - 14 days, or ticarcillin/clavulanate 3.1 grams intravenously every 4 - 6 hours, may be switched to amoxicillin/clavulanate 875 mg by mouth, twice daily, total duration 7 - 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bacterial skin and skin structure infection with a complicating factor, (including a pre-existing skin lesion, or a condition affecting the way the drug gets to the infected area of the body, the body's disease defense (immune) system, or the ability of tissues to heal properly)
* have at least 2 of the following signs and symptoms of skin infection: pain, redness, swelling, hardness, pus formation
* have an infection of one of the following types: wound infections (crush, puncture, cut, gunshot, surgery, bite), infected skin ulcers, or infections in patients with decreased immune system function (HIV infections, diabetes, etc)
* able to provide a sample of tissue from the affected area of the skin

Exclusion Criteria:

* Patients with multiple infected ulcers at separate locations on body
* requiring immediate surgery at the infection site
* having low blood pressure, decreased urination, decreased kidney function, seizure disorder, unstable mental disorder, low white blood cell count, bone infection, shock, or are HIV positive
* having an infection from a bacteria known to be resistant to any of the study drugs
* having a previous allergic or serious reaction to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 1997-01; Study Completion 1998-07 (Actual)

PRIMARY OUTCOMES:
Clinical response rates at post-therapy, categorized as cured, improved, or failed.

SECONDARY OUTCOMES:
Rate of elimination of disease-causing bacteria post-study, by patient, and by bacteria type; Clinical relapse and new infection rates based upon signs and symptoms at post-study; Microbiologic relapse rates

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Graham DR, Talan DA, Nichols RL, Lucasti C, Corrado M, Morgan N, Fowler CL. Once-daily, high-dose levofloxacin versus ticarcillin-clavulanate alone or followed by amoxicillin-clavulanate for complicated skin and skin-structure infections: a randomized, open-label trial. Clin Infect Dis. 2002 Aug 15;35(4):381-9. doi: 10.1086/341026. Epub 2002 Jul 19. PMID 12145720
- See also: A study of the safety and effectiveness of levofloxacin compared to ticarcillin/clavulanate alone or followed by amoxicillin/clavulanate in the treatment of skin infections — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=650&filename=CR005473_CSR.pdf